CLINICAL TRIAL: NCT04672317
Title: A Prospective, Open Clinical Study to Examine the Efficacy and Safety of Neoadjuvant Tislelizumab Combined With Cisplatin-based Chemotherapy in Patients With Locally Advanced Upper Urinary Tract Urothelial Carcinoma
Brief Title: Neoadjuvant PD-1 Monoclonal Antibody Plus Cisplatin-based Chemotherapy in Locally Advanced Upper Tract Urothelial Carcinoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: RenJi Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UTUC-NEOCI
Record Dates: First submitted 2020-12-12; First posted 2020-12-17 (Actual); Last update posted 2020-12-17 (Actual); Status verified 2020-12

CONDITIONS: Neoadjuvant Therapy of Locally Advanced Upper Urinary Tract Urothelial Carcinoma
Keywords: neoadjuvant therapy; radical nephroureterectomy; Tislelizumab; chemotherapy
MeSH Terms: interventions — Drug Therapy

STUDY DESIGN:
Intervention Model Description: Before surgery, patients will receive 2-4 cycles of Tislelizumab (200mg per cycle) in combination with cisplatin-based chemotherapy
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Neoadjuvant arm (Experimental): Patients will receive 2-4 cycles of Tislelizumab (200mg per cycle) in combination with cisplatin-based chemotherapy before radical nephroureterectomy and lymphadenectomy.
  Drug: Tislelizumab 200 mg per cycle, IV on day 14 of every 3-week cycle, for 2-4 cycles prior to radical nephroureterectomy and lymphadenectomy Drug: Cisplatin 70mg/m2 IV on day 2of every 3-week cycle, for 2-4 cycles prior to radical nephroureterectomy and lymphadenectomy. Dose fractionation is permissible.
  Drug: Gemcitabine 1000mg/m2 IV on day 1 and Day 8 of every 3-week cycle, for 2-4 cycles prior to radical nephroureterectomy and lymphadenectomy
  Interventions: Drug: Immunotherapy combined with chemotherapy

INTERVENTIONS:
Drug: Immunotherapy combined with chemotherapy — Patients will receive 2-4 cycles of Tislelizumab (200mg per cycle) in combination with cisplatin-based chemotherapy before radical nephroureterectomy and lymphadenectomy.
  Drug: Tislelizumab 200 mg per cycle, IV on day 14 of every 3-week cycle, for 2-4 cycles prior to radical nephroureterectomy and lymphadenectomy
  Other Names:
  • anti-PD-1 monoclonal antibody Drug: Cisplatin 70mg/m2 IV on day 2of every 3-week cycle, for 2-4 cycles prior to radical nephroureterectomy and lymphadenectomy. Dose fractionation is permissible.
  Drug: Gemcitabine 1000mg/m2 IV on day 1 and Day 8 of every 3-week cycle, for 2-4 cycles prior to radical nephroureterectomy and lymphadenectomy

SUMMARY:
This study is designed prospectively to investigate the safety and efficacy of neoadjuvant PD-1 monoclonal antibody combined with cisplatin-based chemotherapy in patients with locally advanced upper urinary tract urothelial carcinoma (UTUC). Tislelizumab, an anti-programmed death protein-1 (PD-1) monoclonal antibody, was engineered to minimize binding to FcγR on macrophages to abrogate antibody-dependent phagocytosis, a mechanism of T-cell clearance and potential resistance to anti-PD-1 therapy. The safety, tolerability, and efficacy of tislelizumab in patients with PD-L1 positive urothelial carcinoma who progressed during/following platinum-containing therapy was proved in a phase 2 trial (CTR20170071). This trial focuses on the efficacy of Tislelizumab in combination with cisplatin-based chemotherapy to induce pathological down-staging of locally advanced UTUC in neoadjuvant setting.

DETAILED DESCRIPTION:
Neoadjuvant therapy of cisplatin-based chemotherapy has been proved to improve prognosis of muscle invasive UTUC patients in several studies. This study is designed to investigate the safety and efficacy of neoadjuvant PD-1 monoclonal antibody combined with cisplatin-based chemotherapy in patients with locally advanced upper urinary tract urothelial carcinoma (UTUC).

ELIGIBILITY:
Inclusion Criteria:

* 1. Patients that are identified as locally advanced upper urinary tract urothelial carcinoma by ureteroscopic biopsy and imaging diagnosis and are determined as appropriate candidates for radical nephrectomy by an attending urologist; 2. Patients who have a clinical stage of T3-T4, any N, M0 or any T, N1-2, M0; 3. ECOG performance status of 0 to 2; 4. Adequate organ function defined by study-specified laboratory tests;

  1. Hemoglobin ≥90 g/L;
  2. Hematological Absolute neutrophil count (ANC) ≥1.5×109 /L;
  3. Platelets ≥100×109 /L 5. No functional organic disease: T-BIL≤1.5×upper limit of normal (ULN); ALT and AST≤2.5×ULN；eGFR ≥ 60ml/min (MdRD) 6. Agree to comply with scheduled visits, treatment plans, lab tests and any other required study procedures;

Exclusion Criteria:

1. Patients who has received prior therapy of an anti-PD-1, anti-PD-L1, or anti-PD-L2 antibody;
2. Patients who are allergic to monoclonal antibodies or any of its excipients;
3. Patients who have received other anti-tumor treatment (e. g., Steroid therapy, immunotherapy) within 4 weeks or enrolled in other clinical trials;
4. Patients who are pregnant or breastfeeding, or expecting to conceive;
5. Patients who have a known history of Human Immunodeficiency Virus (HIV) (HIV 1/2 antibodies);
6. Patients who have known active Hepatitis B or Hepatitis C;
7. Patients who have active autoimmune disease that has required systemic treatment in the past 2 years;
8. Patients who have received a live vaccine within 30 days prior to the first dose of trial treatment;
9. Patients who have received prior radiation therapy to the bladder;
10. Patients who have bladder cancer;
11. Patients who have received allogeneic hematopoietic stem cell transplantation or solid organ transplantation;
12. Patients who have a history of substance abuse or with a history of mental disorders;
13. Patients who had other malignant tumors in the past five years that have not recovered except for curable tumors that have been cured including basal or squamous skin cancer, localized carcinoma in situ of the cervix or the breast or low-risk prostate cancer, etc;Patients who have active tuberculosis;
14. Patients who have other serious and uncontrollable accompanying diseases that may affect compliance or interfere with the interpretation of results including active opportunistic infections or advanced (severe) infections, uncontrollable diabetes, cardiovascular disease (grade III or IV heart failure defined by the New York Heart Association classification, II degree atrioventricular block and above, myocardial infarction in the past 6 months, unstable arrhythmia or instability angina, cerebral infarction within 3 months, etc.) or lung disease (interstitial pneumonia, history of obstructive lung disease and symptomatic bronchospasm);
15. Patients who have a large amount of pleural fluid or ascites with clinical symptoms or requiring symptomatic treatment.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2020-12-10 (Actual); Primary Completion 2022-06-01 (Estimated); Study Completion 2022-06-01 (Estimated)

PRIMARY OUTCOMES:
Pathological complete response rate | 30 days after surgery
  the absence of visible lesion of carcinoma (ypT0/Tis) and the absence of microscopic lymph node metastases (ypN0) on the final surgical specimen

SECONDARY OUTCOMES:
Pathologic response rate | 30 days after surgery
  The rate of patients that reach pathological downstaging at the time of nephroureterectomy.

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Renji Hospital, Shanghai, Shanghai Municipality, China